CLINICAL TRIAL: NCT03431480
Title: Safety Study of Autologous Cord Blood Stem Cell Treatment in Hypoplastic Left Heart Syndrome Patients Undergoing the Norwood Heart Operation
Brief Title: Safety of Autologous Cord Blood Cells in HLHS Patients During Norwood Heart Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Principal Investigator, Salvatore Pepe, Trial Study Coordinator, Murdoch Childrens Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC37112A
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hypoplastic Left Heart Syndrome; Heart Defects, Congenital; Pediatric Disorder
Keywords: cord blood stem cell; Norwood heart surgery; congenital; heart
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Safety
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hCBMNC (Experimental): Autologous human placental cord blood mononuclear cells (buffy coat fraction)
  Interventions: Biological: Autologous Human Placental Cord Blood Mononuclear Cells

INTERVENTIONS:
Biological: Autologous Human Placental Cord Blood Mononuclear Cells — Autologous human placental cord blood mononuclear cells are infused into the coronary artery during the Norwood heart operation
  Other Names: Cord blood buffycoat mononuclear cells, incl stem cells

SUMMARY:
This study aims to evaluate the safety and feasibility of coronary infusion of autologous placental cord blood mononuclear cells during the Norwood heart operation in newborn hypoplastic left heart syndrome (HLHS) patients.

DETAILED DESCRIPTION:
This is a Phase I, open label safety study. Autologous cord blood mononuclear cells (stem cell containing, cord blood buffy coat fraction) was delivered by coronary infusion during the Norwood cardiopulmonary bypass operation in 10 antenatally diagnosed HLHS patients within 2-3 days of birth. Safety and clinical status monitoring was performed to Stage II surgical intervention for HLHS (at approximately 3 months of age). Treated patients will continue to be assessed beyond the trial during follow up between Stage II and III (Fontan) surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male and females with antenatally diagnosed Hypoplastic Left Heart Syndrome (all types requiring Norwood operation)
* Written informed consent by parents/legal guardian
* Successful aseptic collection of autologous cord blood unit and transfer of buffy coat mononucleocyte fraction to cold storage pending cardiac surgery within 2-4 days

Exclusion Criteria:

Patient:

* does not have autologous cord blood cells available at the time of cardiopulmonary bypass surgery
* has evidence of arrhythmia requiring anti-arrhythmia therapy
* has an additional congenital diagnosis that contributes to conditions such as an immune system disorder, immune deficiency, complex metabolic disorder, brain dysplasia or progressive neurological degenerative disorder
* has other clinical complexity deemed by the cardiac surgeon to make the patient unsuitable for inclusion in the trial

Mother:

• is serum positive for HIV, hepatitis or other significant pathogen and has known allergies to penicillin, streptomycin or other antibiotic

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse cardiac events | 1 month
  Monitoring of adverse events including death, heart or other organ failure, myocardial infarction, sustained/symptomatic ventricular tachycardia, bleeding, stroke

SECONDARY OUTCOMES:
Change in right ventricular function -fractional shortening (% units) | baseline, 1 month, 3 months, 12 months
  Measured by cardiac imaging with serial echocardiography and MRI scans
Change in right ventricular end-diastolic wall thickness (% units) | baseline, 1 month, 3 months, 12 months
  Measured by cardiac imaging with serial echocardiography and MRI scans
Change in right ventricular end-diastolic volume (% units) | baseline, 1 month, 3 months, 12 months
  Measured by cardiac imaging with serial echocardiography and MRI scans
Change in right ventricular end-systolic volume (% units) | baseline, 1 month, 3 months, 12 months
  Measured by cardiac imaging with serial echocardiography and MRI scans
Increase in body weight | baseline, 1 month, 3 months, 12 months
  Body weight measured in kilograms
Composite measure of height and head circumference | baseline, 1 month, 3 months, 12 months
  Body height and head circumference measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Pepe, Principal Investigator — Melbourne Children's Campus (incorporating The Royal Children's Hospital, Murdoch Children's Research Institute, the University of Melbourne Department of Paediatrics); Christian P Brizard, Principal Investigator — Melbourne Children's Campus (incorporating The Royal Children's Hospital, Murdoch Children's Research Institute, the University of Melbourne Department of Paediatrics)
Locations (1):
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be available following study publication and discussion between CIs and other researchers regarding future multicentre studies.

REFERENCES:
- [Derived] Brizard CP, Elwood NJ, Kowalski R, Horton SB, Jones BO, Hutchinson D, Zannino D, Sheridan BJ, Butt W, Cheung MMH, Pepe S. Safety and feasibility of adjunct autologous cord blood stem cell therapy during the Norwood heart operation. J Thorac Cardiovasc Surg. 2023 Dec;166(6):1746-1755. doi: 10.1016/j.jtcvs.2023.07.035. Epub 2023 Jul 30. PMID 37527726